CLINICAL TRIAL: NCT03489577
Title: The Role of Post-traumatic Inhibition of the Innate and Adaptive Immune System in the Development of Infectious Complications in Severely Injured Patients
Acronym: POSEIDON
Status: Terminated | Type: Observational
Why Stopped: Interim analysis provided enough data
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Prof. dr Leenen, Prof. Dr., UMC Utrecht
Other Study IDs: 43279
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Multiple Trauma; Sepsis; Innate Immune Response; Disorder of Neutrophils; Multiple Organ Dysfunction Syndrome
Keywords: Inflammation; Multiple Organ Failure; Sepsis; Wounds and Injuries; Pathologic Processes; Shock; Infection; Systemic Inflammatory Response Syndrome; Neutrophils; PMN; Granulocytes; Innate immunity; ICU; Intensive Care; polytrauma; host-pathogen
MeSH Terms: conditions — Multiple Trauma; Sepsis; Multiple Organ Failure; Inflammation; Wounds and Injuries; Pathologic Processes; Shock; Infections; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients admitted to the Intensive Care Unit after severe injury are prone to suffer from infectious complications and even sepsis. Despite tremendous efforts the etiology of this increased susceptibility to infectious pathogens is incompletely understood. Clinical signs and symptoms as well as current diagnostic clinical tests (WBC, CRP, cytokines, interleukines) lack sensitivity or specificity for adequate prediction of the development of infectious complications or sepsis.

Neutrophil granulocytes, cells of the innate immune system, play an important role in the defence against invading bacterial pathogens and are crucial in preventing fulminant infections. For successful eradication of a bacterium neutrophils need to exert specific functions: chemotaxis, migration, phagocytosis, degranulation and production of radical oxygen species. Much research has focused on the effect of trauma on neutrophil's individual capacities to kill bacteria with conflicting interpretations as a result. For adequate determination of the neutrophil's capacity to eradicate bacteria from tissue of trauma patients we developed novel in-vitro assays in which neutrophils are tested for all of these functions combined. This assay allows us to identify dysfunctional neutrophils adequately.

The main focus of this study is the determination of the functionality of aberrant neutrophils circulating in the peripheral blood of severly injured following trauma.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the ICU
* Expected stay of at least 2 days
* Age: 18 - 80 years
* Informed consent (when proxy consent is obtained and the patient leaves the ICU in good mental health, personal informed consent is additionally necessary)

Exclusion Criteria:

* Immunosuppressive medication
* HIV and related diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma patients likely to be admitted to the intensive care unit of the UMCU
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Bactericidal capacity of neutrophils and sepsis | 15 days following admission on ICU
  The correlation between reduced bactericidal capacity of neutrophils acquired from severely injured patients and the late occurrence of sepsis

SECONDARY OUTCOMES:
Bactericidal capacity of neutrophils and infectious complications | 15 days following admission to the ICU
  The correlation between reduced bacterial killing by neutrophils acquired from trauma patients and the occurrence of infectious complications (e.g pneumonia, meningitis, pericarditis, urinary tract infections, abdominal abscesses)
Bactericidal capacity of neutrophils and pro-inflammatory complications | 15 days following admission to the ICU
  The correlation between bactericidal function of neutrophils and the occurrence of pro-inflammatory complications (SIRS).
Priming capacity of neutrophils and infectious complications | 15 days following admission on the ICU
  The relationship between the responsiveness of neutrophils to a priming stimulus (fMLP) and the occurrence of infectious complications
Complement system and infectious complications | 15 days following admission to the ICU
  The correlation between functionality of the complement system and the occurence of infectious complications.
T-cell proliferation and infectious complications | 15 days following admission on ICU
  The difference in suppression of T-cell proliferation in patients suffering infectious complications versus non-infectious patients.

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Leliefeld, Md, Principal Investigator — UMC Utrecht; Luke PH Leenen, Prof. Dr., Study Chair — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No